CLINICAL TRIAL: NCT00252616
Title: Phase III Study of Early vs. Delayed Goal Enteral Nutrition in Mechanically Ventilated Patients
Brief Title: Timing of Target Enteral Feeding in the Mechanically Ventilated Patient
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Todd Rice, Assistant Professor, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 020744
Record Dates: First submitted 2005-11-09; First posted 2005-11-11 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: Acute Respiratory Failure
Keywords: Mechanical ventilation; acute respiratory failure; early nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): trophic feeds
  Interventions: Behavioral: trophic enteral feeds
- 2 (Active Comparator): Full-calorie feeds
  Interventions: Behavioral: trophic enteral feeds

INTERVENTIONS:
Behavioral: trophic enteral feeds — 10cc/hr

SUMMARY:
This study tests the hypothesis that initial trophic enteral feedings will increase the time alive and free of mechanical ventilation as compared to initial goal enteral feedings in patients who are mechanically ventilated.

DETAILED DESCRIPTION:
Mechanically ventilated patients, within 48 hours of initiating mechanical ventilation, are randomized in a 1:1 fashion to receive trophic enteral feedings for 96 hours followed by advancement to goal feeding rates or initial advancement to goal feeding rates. Primary endpoints are ventilator free days, ICU-free days, gastrointestinal intolerances, development of nosocomial infections, and mortality.

ELIGIBILITY:
Inclusion Criteria: Patients will be eligible for inclusion in the study if they meet the following criteria:

* Mechanical ventilation expected to last at least 72 hours.
* Presence of, or primary physician's intent to place, an enteral feeding tube and begin enteral feeds.

Exclusion Criteria:

* More than 48 hours elapsed since both inclusion criteria met.
* Patient, legal representative, or physician refuses consent or is unavailable to provide consent.
* Patient, legal representative, or physician not committed to full support (Exception: A patient will not be excluded if he/she would receive all supportive care except for attempts at resuscitation from cardiac arrest).
* Presence of malignant or irreversible condition and estimated 28 day mortality greater than 50%.
* Severe or refractory shock.
* Moribund patients not expected to survive 24 hours from start of enteral feeding (as determined by primary medical team).
* Child-Pugh score greater than 10.
* Presence of partial or complete mechanical bowel obstruction, or ischemia, or infarction.
* Current TPN use or intent to use TPN within 7 days.
* Severe malnutrition with BMI less than 18.5 and/or loss of more than 30% total body weight in the previous 6 months.
* Neuromuscular disease impairing the ability to ventilate spontaneously.
* Laparotomy expected within 7 days.
* Unable to raise head of bed 45°.
* greater than 30% total body surface area burns.
* Absence of GI tract/short bowel syndrome - defined as entire length of small bowel totaling 4 feet or less.
* Presence of high-output (> 500 cc/day) enterocutaneous fistula.
* Age less than 13 years
* Allergy to enteral formula

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2003-09; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Ventilator-free days | day 28

SECONDARY OUTCOMES:
ICU-free days | day 28
Mortality | 28 days
Incidence of Gastrointestinal intolerances | day 14
Organ failure-free days | day 28
Changes in inflammation as measured by serum cytokine levels | baseline vs. days 6 and 12
Changes in levels of nutrition as measured by serum albumin, total protein, and pre-albumin | baseline vs. days 6 or 12

CONTACTS AND LOCATIONS:
Overall Officials: Todd W Rice, MD, MSc, Principal Investigator — Vanderbilt University School of Medicine
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Rice TW, Mogan S, Hays MA, Bernard GR, Jensen GL, Wheeler AP. Randomized trial of initial trophic versus full-energy enteral nutrition in mechanically ventilated patients with acute respiratory failure. Crit Care Med. 2011 May;39(5):967-74. doi: 10.1097/CCM.0b013e31820a905a. PMID 21242788